CLINICAL TRIAL: NCT04084626
Title: A Clinical Trial of Programmed Cell Death Protein 1(PD1) Antibody and Lenalidomide as a Treatment for Epstein-Barr Virus-associated Hemophagocytic Lymphohistiocytosis or Chronic Active EBV Infection(CAEBV)
Brief Title: PD1 Antibody and Lenalidomide as a Treatment for EBV-HLH or CAEBV
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, Principal Investigator, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD-1 antibody-EBV
Record Dates: First submitted 2019-09-08; First posted 2019-09-10 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: EBV Infection
MeSH Terms: conditions — Epstein-Barr Virus Infections | interventions — spartalizumab; Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 antibody (Experimental): PD-1 antibody and lenalidomide administered in 2 week cycles for 6 cycles.
  Interventions: Drug: PD1 antibody; Drug: lenalidomide

INTERVENTIONS:
Drug: PD1 antibody — 2mg/kg ivgtt on day 1(age<18 years); 200mg ivgtt on day 1(age >=18 years).
Drug: lenalidomide — 5mg orally once a day（age<18years) ,day 1-14; 10mg orally once a day(age>=18years), day 1-14.

SUMMARY:
The present study was a prospective one-arm clinical study, in which EBV-HLH/chronic active EBV infection patients were selected as the main subjects to evaluate the effect of PD-1 antibody and lenalidomide regimens on ebv-dna and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CAEBV confirmed by 2016 Revised World Health Organization classification.
2. If the patient has previously suffered CAEBV-HLH, the HLH should be in remission.
3. A woman of childbearing age must be determined not to be pregnant by a pregnancy test and is willing to take effective measures to prevent pregnancy during the trial period and ≥12 months after the last administration of the drug; All male subjects used contraceptive methods during the study period and ≥6 months after the last administration;
4. Ages Eligible for Study: 1 Year to 65 Years.
5. Sign the informed consent.

Exclusion Criteria:

1. Heart function above grade II (NYHA).
2. Pregnancy or lactating Women.
3. Allergic to PD-1 antibody or lenalidomide.
4. Active bleeding of the internal organs.
5. uncontrollable infection.
6. Participate in other clinical research at the same time.

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-09-15 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Response rate | 6 months
  The rate of decline in EBV-DNA copy (defined as a 2log decrease in EBV-DNA copy) or negative rate in peripheral blood mononuclear cells and plasma

SECONDARY OUTCOMES:
Spleen size | 6 months
  ultrasonic spleen size
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | through study completion, an average of 1 years
  Adverse events including thyroid function， liver function damage, myelosuppression, infection, bleeding and so on.
survival | 1 year
  from the date of inclusion to date of death, irrespective of cause Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No